CLINICAL TRIAL: NCT00864578
Title: Effects of the Oral Administration of an Association of Forskolin With Rutin and Vitamins B on Intraocular Pressure (IOP) in Patients Affected by Primary Open Angle Glaucoma (POAG) Under Maximun Tolerated Medical Therapy (MTMT)
Brief Title: Effects of Forskolin on Intraocular Pressure in Glaucomatous Patients Under Maximum Tolerated Medical Therapy
Status: Withdrawn | Type: Observational
Why Stopped: loss of interest before enrolment started
Sponsor: Sooft Italia (Industry)
Responsible Party: Prof. MICHELE VETRUGNO, OPHTHALMOLOGY DPT, UNIVERSITY OF BARI (ITALY)
Other Study IDs: KRONEK-MTMT; KRONEK-001
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Primary Open Angle Glaucoma; Intraocular Pressure
Keywords: POAG; IOP; Forskolin; Food supplement
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Elevated intraocular pressure is still the main risk factor for development and progression of glaucoma. Several drugs exist on the market that may decrease IOP in glaucomatous patients. However, some patients cannot reach the target pressure despite a multitherapy with a combination of drugs, and are therefore addressed to surgical treatments. Forskolin is a natural compound that is a receptor-independent adenyl-cyclase activator, that increases intracellular cAMP. It has been shown to be able to decrease IOP after topical application, by a mechanism that is not used by the other drugs. Aim of the present study is to see whether a food supplement containing forskolin (KRONEK) has any effect on the IOP of POAG patients that cannot reach their target pressure, and are therefore on the waiting list for surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-70 Years
* Sex: both
* Pathology: POAG
* Characteristics: Target pressure not achieved with current treatments

Exclusion Criteria:

* Concomitant ocular pathologies
* Previous ocular surgery
* Known hypersensitivity to any of the components in the KRONEK tablets
* Concomitant participation in other trials

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by POAG and already under observation in the centers that take part in this study
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Enrollment, 1, 2, 3, 4 weeks after initiation of treatment

SECONDARY OUTCOMES:
Intraocular pressure fluctuations during the day | Enrollment, 1, 2, 3, 4 weeks after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vetrugno, MD, Principal Investigator — Ophthalmology Dpt., University of Bari, Italy
Locations (1):
- Ophthalmology Department of the University Clinic, Bari, Italy

REFERENCES:
- [Background] Caprioli J, Sears M. The adenylate cyclase receptor complex and aqueous humor formation. Yale J Biol Med. 1984 May-Jun;57(3):283-300. PMID 6093393
- [Background] Daly JW. Forskolin, adenylate cyclase, and cell physiology: an overview. Adv Cyclic Nucleotide Protein Phosphorylation Res. 1984;17:81-9. PMID 6328947
- [Background] Caprioli J, Sears M. Forskolin lowers intraocular pressure in rabbits, monkeys, and man. Lancet. 1983 Apr 30;1(8331):958-60. doi: 10.1016/s0140-6736(83)92084-6. PMID 6132271
- [Background] Lee PY, Podos SM, Serle JB, Camras CB, Severin CH. Intraocular pressure effects of multiple doses of drugs applied to glaucomatous monkey eyes. Arch Ophthalmol. 1987 Feb;105(2):249-52. doi: 10.1001/archopht.1987.01060020103038. PMID 3813959